CLINICAL TRIAL: NCT02544568
Title: Effects of Standardized Meals With Different Compositions of Fat, Protein and Carbohydrate on the Metabolic, Hormonal and Inflammatory Responses in Human
Brief Title: Effects of Standardized Meals on the Metabolic, Hormonal and Inflammatory Responses in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Neda Rajamand Ekberg, M.D/Ph.D, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2007/801-32
Record Dates: First submitted 2015-08-26; First posted 2015-09-09 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus
Keywords: high fat; high protein; high carbohydrate; insulin; glucose
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High-Carb Meal (Experimental): The 3 Groups (Control, T1DM, T2DM) will receive 4 meals with different compositions at 4 occasions (High-Carb, High-Fat, High-Protein, High-Fibr) .
  Interventions: Other: Meals
- High-Protein Meal (Experimental): The 3 Groups (Control, T1DM, T2DM) will receive 4 meals with different compositions at 4 occasions (High-Carb, High-Fat, High-Protein, High-Fibr) .
  Interventions: Other: Meals
- High-Fat Meal (Experimental): The 3 Groups (Control, T1DM, T2DM) will receive 4 meals with different compositions at 4 occasions (High-Carb, High-Fat, High-Protein, High-Fibr) .
  Interventions: Other: Meals
- High-Fibre Meal (Experimental): The 3 Groups (Control, T1DM, T2DM) will receive 4 meals with different compositions at 4 occasions (High-Carb, High-Fat, High-Protein, High-Fibr).
  Interventions: Other: Meals

INTERVENTIONS:
Other: Meals — At 4 different occasions the participants will receive meals with the same amount of calories and different composition of fat, protein, carbohydrate and fiber.The composition of the meals is: Low-fat / high-carbohydrate meal (18 E% proteins, 28 E% fat and 54% carbohydrates), high-fat meal (18 E% protein, 50 E% fat and 31 E% carbohydrate), high-protein meal (40 E% protein, 30 E% fat and 30 E% carbohydrates) and low-fat / high-carbohydrate and high fiber (18 E% proteins, 28 E% fat and 54 E% carbohydrates and 15 gram of fibers).

SUMMARY:
Meal composition is important for blood sugar levels in patients with diabetes. The aim of this study is to investigate if a meal composition of fat, protein and carbohydrate is important for the hormonal and inflammatory responses Patients with type 1 and type 2 diabetes and healthy controls will be included in the study. At four different occasions the participants will receive lunch with the same amount of calories but different composition of fat, protein, carbohydrate and fiber. Blood samples will be taken before and after the meals. The participants will estimate their satiety. In addition participant will fill in questionnaires about their food habits and wellbeing.

This study is the first study to compare both hormonal and inflammatory responses, as well as psychological aspect of the meals, after meals with different composition. Results from this study will help to make recommendation about meal composition which is beneficial for patients with diabetes type 1 and type 2.

DETAILED DESCRIPTION:
Food is an important part of human beings life. During most part of human beings history the shortage of food has been a problem. Today the shortage of food is unknown phenomena in the industrial countries. Instead human being is facing a challenge in obesity epidemic. The number of obese persons has increased since 1980 in all industrial countries. Today only 20 - 25 % of the population in the US has a normal body mass index (BMI). The populations in Europe and Asia are following the same trend. It is known that increased waist (in women > 80 cm and in men > 94 cm) are correlated to insulin resistance, especially in liver because of increased hepatic fat storage. Increased prevalence of obese persons is followed by increased prevalence of patients with impaired glucose tolerance with increased risk for diabetes type 2, cardiovascular disease and cancer.

It is known that impaired glucose tolerance and diabetes type 2 can be prevented efficiently with weight loss, reduced total intake of fat and carbohydrate, increased intake of fiber and physical activity. Three popular diets, 1) low fat, 2) low carbohydrate (high-protein and high-fat) and 3) low glycemic load, have recently received much attention. Long term studies of these different diets have shown inconsistent results. There is a discussion today if a better metabolic control is achieved with low-carbohydrate diet compared to low-fat diet in patients with diabetes type 2 compared to the diet recommended by Swedish National Food Administration. In regards of dietary composition, hyperglycemia and dyslipidemia is determined by the amount and quality of ingested carbohydrates and dietary fats. It has been suggested that postprandial hyperglycemia and hypertriglyceridemia triggers oxidative stress and causes inflammation, metabolic alterations associated with endothelial dysfunction.

An important aspect of satisfaction after a meal is the feeling of satiety. Subjective feelings of hunger are also obviously related to initiation of food behaviors such as intake of snacks. Neophobia, the fear of new or unfamiliar foods, can also be related to the success or failure of food related behavior change. These feelings of satiety are in turn related to factors such as blood glucose levels. Thus the effect of ingested macronutrients on the postprandial glycemic response is one potential mechanism by which foods may affect satiety. Compared to fats and proteins, dietary carbohydrates may have the greatest effect on postprandial glycemia and insulinemia, and may therefore elicit greater appetitive ratings several hours after consumption compared to lower-glycemic meals. Lately some neuroendocrine hormones (ghrelin, resistin etc) and adipokines (leptin and adiponectin) have received attention as regulators of satiety and plausible causes of obesity. The effect of high-fat, high-protein or low-carbohydrate meals on these hormones are not known.

The adverse effects of factors such as chronic stress and depression on general health have been documented for many decades. Apart from having an influence on specific health behaviors, other interacting influences such as general life stress appear to be related directly to alterations in pro-inflammatory and hemostasis processes. The physiological pathways by which psychosocial factors might exert both positive and negative effects on health are numerous and incompletely understood. However, examples of particular interest are findings that suggest that even in relatively healthy persons, chronic negative appraisals of minor life events (hassles) are associated with increased circulating levels of inflammatory factors, whereas persistent positive appraisals of minor life events (uplifts) are associated with decreased levels of such factors. It is thus important to consider general Quality of Life, as well as food-related quality of life together with health and taste attitudes and nutritional knowledge.

Finally the gender aspect is also of importance. Previously it has been presumed that the inflammatory and hormonal responses to different diets are the same in men and women. There are known biological and hormonal differences between men and women. One may question why women get heart infarction later in life compared to men and if the risk factors including inflammatory responses, cholesterol levels and other hormonal changes after different diets are the same in men and women.

The aim of this study is to compare the high-fat, high-protein and low-carbohydrate meal regarding post prandial glucose and triglycerides concentrations in blood as well as the fast inflammatory response, oxidative stress and appetite regulating hormones in healthy subjects and patients with diabetes. Gender differences will be investigated. In general this study will provide information on which meal compositions that are beneficial for patients with diabetes and healthy subjects. Another aim of this study is to investigate if the psychosocial aspect of the meal such as health locus of control, neophobia, satiety and food related Quality of Life is important for the hormonal responses after the meals.

Hypothesis :

1. Meal with high concentration of fiber (15 g) is beneficial for metabolic control in patients with diabetes.
2. Low-carbohydrate meal is beneficial for the metabolic control in patients with diabetes.
3. High-fat meal results in hyperlipidemia which worsens hepatic insulin sensitivity and increases the oxidative stress.
4. High-protein and high-fat meal give earlier satiety and lower blood sugar levels compared to high carbohydrate diet.
5. The perception of the meal affects the metabolic control.

Design:

30 patients with type 1 (T1DM) and 30 patients with type 2 diabetes (T2DM)and 30 healthy Controls (HC) will be included in the study. At four different occasions the participants will eat lunch with different composition of fat, protein, carbohydrate and fiber. All groups are divided in subgroups of men and women. Healthy subjects will receive an oral glucose tolerance test before they are included in the study.

The composition of the meals is: Low-fat / high-carbohydrate meal (18 Eenergi % (E%) proteins, 28 E% fat and 54% carbohydrates), high-fat meal (18 E% protein, 50 E% fat and 31 E% carbohydrate), high-protein meal (40 E% protein, 30 E% fat and 30 E% carbohydrates) and low-fat / high-carbohydrate and high fiber (18 E% proteins, 28 E% fat and 54% carbohydrates and 15 gram of fibers).

Before the study and before the last meal we will measure the waist/hip ratio, BMI and body composition (Bioimpedance). Before the study the participant will document their daily meals during three days. Patients with diabetes should at the same time also document their blood sugar levels (7 times per day, fasting levels, levels before and 2 hours after lunch and dinner and before they go to sleep). Before the other occasions patients will measure their blood sugar levels during one day (7 times).

The participants will eat a standardized breakfast at home in the morning before participating in the study. They will eat one of following meals as lunch at 11:30 am: a low-fat and high-carbohydrate diet recommended by Swedish National Food Administration, a high-protein meal, a high-fat meal or a low-fat and high-carbohydrate diet with 15 g of fibers. At each occasions blood samples will be taken 30 minutes and 5 minutes before the lunch and on 30-minute intervals for the following four hours after the lunch. The blood samples will be analysed for hormones regulating blood sugar levels, appetite regulating hormones, marker of oxidative stress and markers of inflammation and endothelia dysfunctions. We have previously shown that insulin sensitivity in liver can be estimated measuring Insulin like Growh factor- I (IGF-I) and Insulin like Growth Factor Binding Protein-1 (IGFBP-1). These hormones will be analyzed in blood samples.

The participants will estimate their satiety and their desire to eat in parallel at the time blood samples are withdrawn. At each occasion participants will fill in forms about their general perception of the food and how they estimate their own health.

In case a participant do not follow throughout the whole study the results will be analyzed and used in group wise comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 1 DM (age 20-75 years)
* Patient with type 2 DM (diabetes duration more than 5 years, age 20- 75 years, BMI 26 - 33 kg/m2).
* Healthy volunteers (age 20- 75 years).

Exclusion Criteria:

* Heart failure - the New York Heart Association (NYHA) Functional Classification III-IV
* Kidney failure - S-Creatinin mora than 200 micromol/L
* Liver disease - Alanine aminotransferase (ALAT) more than 2 mikroKat/L

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration [Cmax] of glucose and triglycerides | 1 year
  The maximum plasma concentration of glucose and triglyceres after the meals

SECONDARY OUTCOMES:
Maximum plasma concentration [Cmax] of IGFBP-1 | 2 year
  The maximum plasma concentration of IGFBP-1 after the meals
Maximum plasma concentration [Cmax] of marker of oxidative stress | 2 year
  The maximum plasma concentration of markers of oxidative stress after the meals
Maximum plasma concentration [Cmax] of inflammatory markers | 2 year
  The maximum plasma concentration of inflammatory markers after the meals
Maximum plasma concentration [Cmax] of appetite regulatory hormones | 2 years
  The maximum plasma concentration of apetite regulatory hormones after the meals
Maximum plasma concentration [Cmax] of glucagon | 2 years
  The maximum plasma concentration of glucagon after the meals

CONTACTS AND LOCATIONS:
Overall Officials: Neda R Ekberg, M.D./Ph.D., Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden